CLINICAL TRIAL: NCT01661335
Title: Efficacy of Aprepitant (Emend®) in Children Receiving Highly Emetogenic Chemotherapy
Brief Title: Efficacy of Aprepitant (Emend®) in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 0413
Record Dates: First submitted 2012-06-18; First posted 2012-08-09 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Nausea; Vomiting; Childhood Cancer
Keywords: Nausea; Vomiting; Children; Aprepitant; Emend®
MeSH Terms: conditions — Nausea; Vomiting; Neoplasms | interventions — Ondansetron; Dexamethasone; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ondansetron, dexamethasone, aprepitant (Experimental): Arm A: Ondansetron 0.15 mg/kg (max 16 mg) IV or PO every 8 hours for at least 3 days, but no longer than 5 days; dexamethasone 0.2mg/kg (max 10 mg) IV or PO daily for at least 3 days, but no longer than 5 days; and aprepitant 3 mg/kg (max 125 mg) PO on day 1, and aprepitant 2 mg/kg (max 80 mg) PO on days 2 and 3 during the first investigational antiemetic cycle. During the next investigational antiemetic cycle, members of this arm will be crossed-over into the placebo arm, where the aprepitant will be replaced by placebo and the dexamethasone dose will be increased to 0.4 mg/kg (max 20 mg) daily.
  Interventions: Drug: Ondansetron, dexamethasone, aprepitant
- Ondansetron, Dexamethasone, placebo (Placebo Comparator): Arm B: Ondansetron 0.15 mg/kg (max 16 mg) IV or PO every 8 hours for at least 3 days, but no more than 5 days; dexamethasone 0.4 mg/kg (max 20 mg) IV or PO daily for at least 3 days, but no more than 5 days; and a PO placebo for 3 days during the first investigational antiemetic cycle. During the second cycle, members this group will be crossed-over to the experimental arm, where the placebo will be replaced by aprepitant and the dexamethasone will be decreased by 50%.
  Interventions: Drug: Ondansetron, Dexamethasone, placebo

INTERVENTIONS:
Drug: Ondansetron, dexamethasone, aprepitant — Ondansetron 0.15 mg/kg (max 16 mg) IV or PO every 8 hours for at least 3 days, but no longer than 5 days; dexamethasone 0.2mg/kg (max 10 mg) IV or PO daily for at least 3 days, but no longer than 5 days; and aprepitant 3 mg/kg (max 125 mg) PO on day 1, and aprepitant 2 mg/kg (max 80 mg) PO on days 2 and 3 during the first investigational antiemetic cycle. During the next investigational antiemetic cycle, members of this arm will be crossed-over into the placebo arm, where the aprepitant will be replaced by placebo and the dexamethasone dose will be increased to 0.4 mg/kg (max 20 mg) daily.
  Other Names: Aprepitant = Emend; ARM A
  Arms: Ondansetron, dexamethasone, aprepitant
Drug: Ondansetron, Dexamethasone, placebo — Ondansetron 0.15 mg/kg (max 16 mg) IV or PO every 8 hours for at least 3 days, but no more than 5 days; dexamethasone 0.4 mg/kg (max 20 mg) IV or PO daily for at least 3 days, but no more than 5 days; and a PO placebo for 3 days during the first investigational antiemetic cycle. During the second cycle, members this group will be crossed-over to the experimental arm, where the placebo will be replaced by aprepitant and the dexamethasone will be decreased by 50%.
  Other Names: ARM B
  Arms: Ondansetron, Dexamethasone, placebo

SUMMARY:
The purpose of this study is to find out whether or not adding aprepitant(Emend®) to the standard therapy will help children who receive chemotherapy to have less nausea and vomiting.

DETAILED DESCRIPTION:
1.1 Primary Aim To determine the efficacy of aprepitant (Emend®) in preventing and reducing chemotherapy-induced nausea and vomiting (CINV) when added to standard antiemetic drug regimens for children receiving highly emetogenic chemotherapy. The working hypothesis will be that standard therapy + aprepitant is superior at preventing CINV than standard therapy + placebo.

1.2 Secondary Aim To evaluate the safety and toxicity of aprepitant (Emend®) in children receiving highly emetogenic chemotherapy when compared to standard antiemetic therapy + placebo.

ELIGIBILITY:
Inclusion Criteria:

under 20.99 years of age at enrollment

Scheduled to receive two identical cycles of highly emetogenic[1] chemotherapy for treatment of a primary malignancy, including:

Chemotherapy with any one or more of the following single agents in any combination:

* Carboplatin
* Carmustine >250 mg/m2
* Cisplatin
* Cyclophosphamide ≥1 g/m2
* Dactinomycin
* High dose Methotrexate ≥ 5 g/m2

Or any of the following defined combinations:

* Cyclophosphamide + anthracycline
* Cyclophosphamide + etoposide
* Cytarabine 150-200 mg/m2 + daunorubicin
* Cytarabine 300 mg/m2 + etoposide
* Cytarabine 300 mg/m2 + teniposide
* Doxorubicin + ifosfamide
* Doxorubicin + methotrexate 5 g/m2
* Etoposide + ifosfamide

Exclusion Criteria:

* Patients who have received aprepitant in the past.
* Patients who demonstrate evidence of increased intracranial pressure.

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Efficacy of aprepitant (Emend®) measured through a complete response | Up to 11 weeks, or until 3 weeks after the second course of the study regimen
  • Percentage of study subjects who demonstrate a complete response, defined as no episodes of emesis and no use of rescue medications during the investigational antiemetic cycles.
Efficacy of aprepitant (Emend®) measured through episodes of emesis and use of rescue medication. | Up to 11 weeks, or until 3 weeks after the second course of the study regimen
  * The total episodes of emesis within 7 days of the first chemotherapy administration of each cycle.
  * The total number of administrations of rescue medications given for breakthrough nausea or vomiting.
Efficacy of aprepitant (Emend®) measured through impact of chemotherapy induced nausea and vomiting on daily life | Up to 11 weeks, or until 3 weeks after the second course of the study regimen
  • A modified, 5-day recall version of the Functional Living Index-Emesis (FLIE) questionnaire
Efficacy of aprepitant (Emend®) measured through a pictorial nausea scale | Up to 11 weeks, or until 3 weeks after the second course of the study regimen
  • A modified version of the Baxter Animated Retching Faces (BARF) scale, administered daily.

SECONDARY OUTCOMES:
Safety of aprepitant (Emend®) | Up to 11 weeks, or until 3 weeks after the second course of the study regimen
  * Occurrence of adverse events as per the NCI Common Terminology Criteria for Adverse Events (CTCAE) v.4.0. These will be reported spontaneously or on inquiry by the investigator/study nurse, and continuously monitored throughout the trial.
  * Weekly complete blood count (CBC) for 3 weeks after each investigational antiemetic cycle.
  * Weekly complete metabolic profile (CMP) for 3 weeks after each investigational antiemetic cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Rene McNall-Knapp, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Jimmy Everest Center for Cancer and Blood Disorders in Children, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No